CLINICAL TRIAL: NCT03811210
Title: Using the Norm Range to Predict the Effect of Food Portion Size Reductions on Compensation
Brief Title: Using the Norm Range to Predict the Effect of Food Portion Size Reductions on Compensation Over 5 Days
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Principal Investigator, Eric Robinson, Reader in Psychological Sciences, University of Liverpool
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Portion size trial
Record Dates: First submitted 2019-01-17; First posted 2019-01-22 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Portion Size
MeSH Terms: interventions — Portion Size

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: portion size — Smaller than normal portion size - the intervention is the main meal component size perceived as 'smaller than normal' that participants are provided with during lunch and dinner in the laboratory.
  Small-normal portion size - the intervention is the main meal component size perceived as 'small-normal' that participants are provided with during lunch and dinner in the laboratory.
  Large-normal portion size - the intervention is the main meal component size perceived as 'large-normal' that participants are provided with during lunch and dinner in the laboratory.

SUMMARY:
Reducing food portion size is a potential strategy to reduce energy intake. However it is unclear at what point consumers compensate for reductions in portion size by increasing energy intake from other items. This could result in no overall benefit of reducing food portion sizes. The investigators tested the hypothesis that reductions to the portion size of components of a main meal will only result in significant compensatory eating when the reduced portion size is no longer visually perceived as 'normal'. In a crossover experiment, participants were served different sized portions during lunch and dinner over 5 days: a 'large-normal', a 'small-normal', and a 'smaller than normal' portion. Intake from all other meal components consumed in the laboratory were measured.

ELIGIBILITY:
Inclusion Criteria:

* willing to consume the test foods
* BMI between 22.5 - 32.5

Exclusion Criteria:

* food allergies, intolerances or specific dietary requirements (including being vegetarian or vegan)
* history of eating disorders
* taking medication which affected appetite
* participated in a portion size studies in the past 12 months, or in dieting or weight loss trials in the past 4 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2018-12-07 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Acute compensatory energy intake | Immediate (within single meal occasion)
  Energy intake from main meal components that are not varied by portion size
Total meal energy intake | Immediate (within single meal occasion)
  Energy intake from all main meal components (including those that are and are not varied by portion size)
Total daily energy intake | Over 5 x full days
  Energy intake from all foods consumed, including those provided in the laboratory and those self-reported

SECONDARY OUTCOMES:
Moderate-vigorous physical activity | Over 5 x full days
  Moderate-vigorous physical activity (recorded using accelerometer device)
Discretionary Leisure-time physical activity | Over 5 x full days
  Discretionary Leisure-time physical activity (recorded with self-report measure International Physical Activity Questionnaire)
Appetite | Over 5 x full days (measured before and after each meal occasion)
  Hunger and fullness sensations before and after laboratory-based meals (self-reported on visual analog scales anchored at 0 'not at all' to 100 'extremely')

CONTACTS AND LOCATIONS:
Locations (1):
- Ashleigh Haynes, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for primary outcome measures, demographic variables, and data reported in resulting publication will be made freely available on Open Science Framework
Supporting Information: Study Protocol, SAP
Time Frame: Study protocol and statistical analysis plan, along with IPD data will be made publicly available on Open Science Framework when results are published
Access Criteria: Data will be freely accessible.

REFERENCES:
- [Derived] Haynes A, Hardman CA, Halford JCG, Jebb SA, Mead BR, Robinson E. Reductions to main meal portion sizes reduce daily energy intake regardless of perceived normality of portion size: a 5 day cross-over laboratory experiment. Int J Behav Nutr Phys Act. 2020 Feb 12;17(1):21. doi: 10.1186/s12966-020-0920-4. PMID 32050979